CLINICAL TRIAL: NCT04179045
Title: A Registry Trial of the Bioheart Rapamycin Drug-Eluting Bioresorbable Coronary Stent System in Patients With Coronary Artery Disease: BIOHEART Ⅲ
Brief Title: A Registry Trial of The Bioheart Rapamycin Drug-Eluting Bioresorbable Coronary Stent System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Bio-heart Biological Technology Co., Ltd. (Industry)
Collaborators: CCRF Inc., Beijing, China (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BXA 2019001
Record Dates: First submitted 2019-11-18; First posted 2019-11-26 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Coronary Artery Disease
Keywords: Bioresorbable Vascular Scaffold System; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bioheart (Experimental): Subjects have CAD with one or two de novo native coronary artery lesions and will be treated with Bioheart Rapamycin Drug-Eluting Bioresorbable Coronary Stent System. There will be only one arm in this study.
  Interventions: Device: The Bioheart Rapamycin Drug-Eluting Bioresorbable Coronary Stent System

INTERVENTIONS:
Device: The Bioheart Rapamycin Drug-Eluting Bioresorbable Coronary Stent System — Subjects enrolled will be treated with Bioheart Rapamycin Drug-Eluting Bioresorbable Coronary Stent.

SUMMARY:
This study is a prospective, multi-center single arm registry trial, planning to enroll 785 subjects. All subjects will receive clinical follow-up at 1 month, 6 month, 9 month and 1, 2, 3, 4, 5 year after index procedure. The primary endpoint will be target lesion failure (TLF) at 1 year after index procedure,which will be analyzed to evaluate the efficacy and safety of the device.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria:

1. Age from 18 to 75 years old, man or non-pregnant woman.
2. Subjects with asymptomatic ischemic evidence, stable or unstable angina, or old myocardial infarction, are suitable for selective PCI.
3. Subjects without contraindications of coronary artery bypass grafting (CABG).
4. Subjects are able to understand the purpose of this study, volunteer to participate and sign informed consent.

Angiographic Inclusion Criteria:

1. One or two de novo target lesions

   1. If subject has only one target lesion, the second non-target lesion must be treated but the non-target lesion must be present in a different epicardial vessel; the non target lesion must be treated first and successfully prior to the subjects' register.
   2. If there are two target lesions, they must be present in different epicardial vessels.
   3. The definition of epicardial vessels means the left anterior descending artery (LAD), the left circumflex artery (LCX), and the right coronary artery (RCA) and their branches. Thus, for example, the subject must not have lesions requiring treatment in both the LAD and a branch.
2. Target lesion diameter stenosis is estimated visually ≥ 70% (or ≥ 50% with clinical evidence of myocardial ischemia), with TIMI flow grade ≥1; Target lesion length ≤24mm (visually); target lesion diameter between ≥2.5 mm to ≤ 4.00 mm.
3. Each target lesion must be covered completely by one scaffold.

Exclusion Criteria:

General Exclusion Criteria:

1. Any newly onset acute myocardial infarction within 1 week or, myocardial enzymes does not return to normal level after myocardial infarction.
2. Target vessel has been implanted with stents within 1 year before procedure.
3. Subjects with severe heart failure (≥ grade III NYHA) or left ventricular ejection fraction <35% (accessed by ultrasound or left ventricular angiography).
4. subject with severe kidney functional damaged before procedure: serum creatinine>2.0mg /dl (176.8μmol / L) or subject is receiving hemodialysis.
5. Subjects with high bleeding risk, with active gastrointestinal ulcers, history of cerebral hemorrhage or history of subarachnoid hemorrhage, history of ischemic stroke within the past six months, with contraindications of anti-platelet agents and anticoagulants, and subjects cannot receive antithrombolytic therapy.
6. subject is known hypersensitive or allergic to aspirin, clopidogrel, heparin, contrast agent, polylactic acid polymer and rapamycin.
7. The subject's life expectancy is less than 24 months.
8. Subjects is currently participating in other drug or medical device clinical trial that has not yet completed its primary endpoint .
9. Subjects have received any solid organ transplants or are ready to undergo organ transplant.
10. Subjects have unstable arrhythmia, such as high-risk ventricular premature beats, and ventricular tachycardia.
11. Subjects receive chemotherapy for tumor.
12. Subjects have received or planning to receive coronary or chest radiotherapy.
13. Subjects with Immunosuppressive, autoimmune diseases, have planned to receive or underwent immunosuppressive therapy.
14. Subjects have planned to receive or are receiving long-term anticoagulation therapy, such as heparin, warfarin and so on.
15. Subjects have planned to receive selective surgery within 6 months, which requires them to discontinue aspirin or clopidogrel.
16. Blood tests showed that the platelet count is less than 100 × 10^9 / L, or more than 700 × 10^9 / L, the white blood cells count is less than 3 × 10^9 /L.
17. subject with diagnosed or suspected liver cirrhosis.
18. Subjects with diffuse peripheral vascular disease, that precludes safe 6 French sheath insertion.

Angiographic exclusion criteria:

These exclusion criteria apply to the target or non-target lesion(s), target or non-target vessel(s):

1. Target or non-target lesion(s) located in left main.
2. Subjects with triple vessel lesion in LAD, LCX or RCA, which all need to be treated.

These exclusion criteria apply to the target lesion(s) or target vessel(s):

1. Target lesion located in left main.
2. Target lesion located in the aorto-ostial of RCA (within 3 mm of the origin of the RCA).
3. Target lesion located within 3 mm of the origin of the LAD and LCX.
4. Lesion involving a bifurcation with a:

   1. Side branch ≥ 2.5 mm in diameter, or
   2. Side branch with diameter stenosis ≥ 50%, or
   3. Side branch requiring protection guide wire, or
   4. Side branch requiring pre-dilatation.
5. Anatomy proximal to or within the lesion that may affect delivery of the Bioheart, including:

   1. Extreme angulation (≥ 90°) proximal to or within the target lesion, or
   2. Excessive tortuosity (≥ two 45° angles) proximal to or within the target lesion, or
   3. Moderate or heavy calcification proximal to or within the target lesion.
6. Target lesion involves a myocardial bridge.
7. Target vessel contains thrombus as indicated in the angiographic images or IVUS.
8. Prior to the index procedure target vessel has been previously treated with a stent at any time such that the Bioheart stent would need to cross the stent to reach the target lesion.
9. Target vessel has been previously treated with a stent and the target lesion is within 5 mm proximal to a previously treated lesion.
10. Target lesion cannot meet the following outcomes, after the complete balloon pre-dilatation:

    1. Residual (DS %) is < 40% (per visual estimation), ≤ 20% is strongly recommended;
    2. TIMI Grade-3 flow (per visual estimation);
    3. No angiographic complications (e.g., no-reflow, distal embolization, side branch closure)
    4. No dissections NHLBI grade D-F;
    5. No chest pain lasting > 5 minutes, and;
    6. No ST depression or elevation lasting > 5 minutes.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 785 (Estimated)
Dates: Start 2021-03-01 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
TLF | 1 year after index procedure
  Target lesion failure, consists of cardiac death, MI attributed to the target vessel, and ischemic driven - target lesion revascularization (ID-TLR).

SECONDARY OUTCOMES:
The device-oriented composite（DoCE） / TLF | at 1, 6, 9 month and 1, 2, 3, 4, 5 year after index procedure
  consists of cardiac death, MI attributed to the target vessel, and ischemic driven- target lesion revascularization (ID-TLR).
The patient-oriented composite（PoCE） | at 1, 6, 9 month and 1, 2, 3, 4, 5 year after index procedure
  includes all-cause mortality, any MI, and any revascularization. Death（Cardiac death，Vascular death，Non-cardiovascular death）; Myocardial Infarction (target vessel MI, non-target vessel MI); Target lesion Revascularization（ischemic driven, non-ischemic driven） target vessel Revascularization （ischemic driven, non-ischemic driven）; Any Revascularization （ischemic driven, non-ischemic driven）.
Stent Thrombosis（ARC） | at 1, 6, 9 month and 1, 2, 3, 4, 5 year after index procedure
  Timing：Acute, Subacute, Late,Very late stent thrombosis Definite and Probable Stent Thrombosis
Device success | immediately after index procedure
  defined as attainment of residual stenosis less than 30% by visual estimation and TIMI flow grade 3 post stent implantation
Lesion success | immediately after index procedure
  defined as attainment of diameter residual stenosis less than 30% by visual estimation and TIMI flow grade 3, after the target lesion treated by any PCI methods
Clinical success | up to 7 days after index procedure
  defined as attainment of lesion success and without any major adverse cardiac events during hospitalization (up to 7 days after index procedure)

CONTACTS AND LOCATIONS:
Overall Officials: Guosheng Fu, Professor, Principal Investigator — Sir Run Run Shaw Hospital (SRRSH), affiliated with the Zhejiang University School of Medicine
Locations (5):
- China (5):
  - Beijing Anzhen Hospital Capital Medical University, Beijing, Beijing Municipality
  - BeijingChao-YangHospital, Beijing, Beijing Municipality
  - Nanfang Hospital, Guangzhou, Guangdong
  - Taida International Cardioascular Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital (SRRSH), affiliated with the Zhejiang UniversitySchool of Medicine, Hangzhou, Zhejiang